CLINICAL TRIAL: NCT02101684
Title: Open Label Phase II Clinical Trial of Orteronel (TAK-700) in Metastatic or Advanced Non-resectable Granulosa Cell Ovarian Tumors. The Greko II Study.
Brief Title: Orteronel (TAK-700) in Metastatic or Advanced Non-resectable Granulosa Cell Ovarian Tumors. The Greko II Study.
Acronym: Greko II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Grupo Español de Tumores Huérfanos e Infrecuentes (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETHI 2013-01; 2013-003128-35 (EudraCT Number)
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Metastatic or Advanced Non-resectable Granulosa Cell Ovarian Tumors
Keywords: Orteronel, Granulosa Cell Tumour
MeSH Terms: conditions — Neoplasm Metastasis; Granulosa Cell Tumor | interventions — orteronel; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orteronel 300mg b.i.d. (Experimental): Orteronel 300mg BID (600mg per day) will be administered to all included patients in a 28 days cycle schedule.
  Interventions: Drug: Orteronel 300mg BID

INTERVENTIONS:
Drug: Orteronel 300mg BID

SUMMARY:
Granulosa Cell ovarian carcinoma is an infrequent subtype of neoplasia well differentiated from epithelial tumors. They account for 5% of all ovarian malignancies and, with an incidence of 0.4-1.2 cases per 100000 habitants, is considered as a rare disease.

Though most cases are identified at initial stages and can be cured through surgical resection, distant recurrences have been documented even 10 years after resecting the primary tumor. At advanced stage it is a lethal disease.

Unfortunately because of the low incidence of this disease randomized clinical trials are lacking. In fact current evidence for treatment is provided by case reports, retrospective studies and phase II clinical trials performed one decade ago.

Orteronel, a novel, orally active, selective inhibitor of 17,20-lyase, is being developed as an endocrine therapy for relevant hormone-sensitive cancers such as prostate cancer and breast cancer. Orteronel is expected to suppress sex hormone levels in both circulation and relevant hormone-dependent malignant tissue. Since sex hormone overproduction has been demonstrated in granulosa cell ovarian tumors and seems to play a major role in this disease, this study will assess the efficacy or orteronel treating such tumors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent.
* Patients, even if surgically sterilized who:

  1. Agree to practice effective barrier contraception during the entire study treatment period and for 4 months after the last dose of study drug, or
  2. Agree to completely abstain from intercourse.
* Patients 18 years or older.
* Screening clinical laboratory values as specified below:
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be <=2.5 X ULN.
* Total bilirubin <=1.5 X ULN.
* Estimated creatinine clearance using the Cockcroft-Gault formula must be >40 mL/minute.
* Absolute neutrophil count (ANC) >=1500/mcL and platelet count >=100,000/mcL.
* Histologically confirmed granulosa cell ovarian tumor with locally advanced non-resectable or metastatic disease, measurable or evaluable by RECIST.
* Availability of sufficient biopsy material to confirm the malignant diagnosis of granulosa cell ovarian tumor by a centralized pathologist and to perform the determine the FOXL2 402C mutation → G (C134W). However study entry will be allowed based just on the histological local diagnosis.
* Life expectancy >=12 weeks
* Screening calculated ejection fraction of greater than or equal to normal by multiple gated acquisition (MUGA) scan, or by echocardiogram (ECHO).
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before first dose of study drug/randomization.

Exclusion Criteria:

* History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 (NCI CTCAE, version 4.02)(56), thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (eg, pericardial effusion restrictive cardiomyopathy) within 6 months prior to first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
* New York Heart Association Class III or IV heart failure.
* ECG abnormalities of:

  1. Q-wave infarction, unless identified 6 or more months prior to screening
  2. QTc interval > 460 msec
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum ?- human chorionic gonadotropin (?-hCG) pregnancy test result obtained during screening.
* Patient has received other investigational drugs within 28 days before enrollment
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy.
* Prior therapy with orteronel, ketoconazole, abiraterone, aminoglutethimide or enzalutamide.
* Patients received radical radiotherapy <= 4 weeks before starting the study treatment or who have not recovered from the toxicities of radiotherapy. Palliative radiotherapy of painful bone lesions is allowed up to 14 days before the start of study treatment.
* Known hypersensitivity to compounds related to orteronel or to orteronel excipients.
* Uncontrolled hypertension despite appropriate medical therapy (BP of greater than 160 mmHg systolic and 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the Screening visit). Note: patients may be rescreened after adjustment of antihypertensive medications.
* Known active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator?s opinion, potentially interfere with participation in this study.
* Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of orteronel, including difficulty swallowing tablets.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Clinical benefit at 6 months | 6 months
  Clinical benefit is defined as the average of patients with radiological response (partial or complete) plus stable disease longer than 6 months by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Response Rate | Every 8 weeks, during 6 months
  Overall Response Rate according to RECIST 1.1 criteria.
Progression free survival | Every 8 weeks, during 6 months
  Progression Free Survival defined as the time from the administration of the first dose of treatment to disease progression or death from any cause.
Overall Survival | Every 12 weeks, untill death
  Overall Survival defined as the time from first dose of treatment to patient death from any cause
Reduction of sex hormones production. | Every 8 weeks, during 6 months
  Significant reduction of sex hormones production will be considered as at least a reduction to half the basal level confirmed in one determination one month apart.
Toxicity profile | Every 4 weeks, untill end of treatment (6 months estimated)
  Frequency of each adverse event per patient

CONTACTS AND LOCATIONS:
Overall Officials: Jesús García-Donas, MD, Study Director — Hospital Universitario Madrid Sanchinarro; Alicia Hurtado, MD, Principal Investigator — Hospital Universitario Fundación Alcorcón; Juan Cueva, MD, Principal Investigator — COMPLEXO HOSPITALARIO UNIVERSITARIO DE SANTIAGO; Laia Garrigos, MD, Principal Investigator — Hospital del Mar; María Jesús Rubio, MD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL REINA SOFÍA; Andrés Redondo, MD, Principal Investigator — Hospital Universitario La Paz; Isabel Bover, MD, Principal Investigator — Hospital Son Llatzer; Nuria Lainez, MD, Principal Investigator — Complejo Hospitalario de Navarra; Ana Santaballa, MD, Principal Investigator — Hospital Universitario La Fe
Locations (9):
- Spain (9):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Del Mar, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitari I Politècnic La Fe, Valencia

REFERENCES:
- [Derived] Garcia-Donas J, Garrigos L, Lainez N, Santaballa A, Redondo A, Cueva JF, Rubio MJ, Prieto M, Lopez-Guerrero JA, Garcia-Casado Z, Barquin A, Grande E, Alia EG, Sevillano E, Bover I, Grazioso TP, Sanchez-Escribano R, Hurtado A, Navarro P, Rodriguez-Moreno JF. Open-label phase II clinical trial of orteronel (TAK-700) in metastatic or advanced non-resectable granulosa cell ovarian tumors: the Greko II study (GETHI2013-01). Clin Transl Oncol. 2025 Jul;27(7):3223-3231. doi: 10.1007/s12094-024-03827-4. Epub 2024 Dec 30. PMID 39738931